CLINICAL TRIAL: NCT03608683
Title: Evaluation of Open Surgical Treatment of Abdominal Aortic Pathology With Hostile Necks, Para-/Juxra-renal and Sovrarenal Pathology at Short, Mid and Long Term
Brief Title: Evaluation of the Treatment of Abdominal Aortic Pathology With Hostile Necks, Para-/Juxra-renal and Sovrarenal Pathology at Short, Mid and Long Term
Acronym: p-AAA
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Mascia Daniele, Principal Investigator, IRCCS San Raffaele
Other Study IDs: p-AAA
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-02

CONDITIONS: Proximal Abdominal Aortic Aneurysms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although open repair (OR) is currently reported as the gold standard of treatment, fenestrated endovascular repair (FEVAR) is being increasingly applied for the treatment of proximal abdominal aortic aneurysms (p-AAA) such as hostile-necked, juxta-, para- and supra-renal aortic aneurysms.1 Nevertheless, advantages of FEVAR in terms of lowering postoperative complications, should be balanced with the need of both complex device configurations and operators with large endovascular expertise. The aim of this study is to report the experience of Data from patients treated will be prospectively collected. All post-operative results will be recorded. Major adverse event (MAE) are defined as the presence of one of the following: all-cause mortality, bowel ischemia, myocardial infarction, paraplegia, respiratory failure, stroke and renal insufficiency.

Furthermore, the pre-operative contrast-enhanced computed tomography scans (CTA) of all patients, stored in the hospital PACS, will be analyzed on the dedicated workstation with OsiriX software (Pixmeo sarl, Bernex, Switzerland) currently employed in our Unit for imaging assessment.

Patients will undergo standard control with the execution of a Doppler ultrasound and creatinine serum levels at 1, 6, 12, 24, 36, 48 and 60 months. A CTA will also be performed at 12 months as per standard clinical practice.

of p-AAA treatment.

DETAILED DESCRIPTION:
Primary end-point is to evaluate the mortality and major adverse events (MAE) at 30 days, 2 years and 5 years prospectively in the cohort of patients p-AAA treated by means of open repair in the next 100 patients that will be treated between 2018 and 2020 in the Vascular Surgery Unit of the San Raffaele Hospital.

Data from patients treated will be prospectively collected. All post-operative results will be recorded. Major adverse event (MAE) are defined as the presence of one of the following: all-cause mortality, bowel ischemia, myocardial infarction, paraplegia, respiratory failure, stroke and renal insufficiency.

Patients will undergo standard control with the execution of a Doppler ultrasound and creatinine serum levels at 1, 6, 12, 24, 36, 48 and 60 months. A CTA will also be performed at 12 months as per standard clinical practice The 100 patients that will be enrolled until December 2020 will also sign an "ad hoc" consents, specific for this study.

Sensitive patient information will not be available during data analysis. The clinical study will be carried out according to the ethical principles of the Declaration of Helsinki and following the active regulations on observational studies.

Expected results are:

* death at 30 days: 2%
* any MAE at 30 day: 25% Patients characteristics and anatomical data on the visceral vessels will be analyzed on Wizard Statistics software to investigate the presence of statistically significant Pearson correlations among the identified variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years,
* Patient undergoing treatment of p-AAA pathology at San Raffaele Hospital

Exclusion Criteria:

• Incomplete imaging quality not including the arterial segments to be studied (visceral vessels) or with a high slice thickness (> 1.5 mm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aneurysm with hostile, para- / juxta-renal and supra-renal collars, undergoing open or surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Percent of participants mortality and major adverse events (MAE) | until 2025
  valuate the mortality and major adverse events (MAE) at 30 days, 2 years and 5 years prospectively in the cohort of patients p-AAA treated by means of open repair in the next 100 patients that will be treated between 2018 and 2020.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

REFERENCES:
- [Result] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Result] Sugimoto M, Takahashi N, Niimi K, Kodama A, Banno H, Komori K. Long-term fate of renal function after open surgery for juxtarenal and pararenal aortic aneurysm. J Vasc Surg. 2018 Apr;67(4):1042-1050. doi: 10.1016/j.jvs.2017.07.121. Epub 2017 Sep 28. PMID 28964618